CLINICAL TRIAL: NCT04618601
Title: Diuretic and Natriuretic Effect of High-dose Spironolactone in Patients With Acute Heart Failure
Acronym: DANAUS-AHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Chris Kapelios, Cardiology Fellow, Laikο General Hospital, Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15606
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure Acute; Heart Failure; With Decompensation
Keywords: diuretic resistance; spironolactone; cardio-renal syndrome; diuretics; natriuresis; heart failure
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose spironolactone (Active Comparator): Participants in this arm will receive high doses of per os spironolactone, defined as doses ≥100 mg daily, on top of standard of care treatment for acute heart failure
  Interventions: Drug: Spironolactone
- Standard of care (No Intervention): Participants in this arm will standard of care treatment for acute heart failure, which may include per os spironolactone at a maximum dose of 50 mg daily

INTERVENTIONS:
Drug: Spironolactone — Patients randomized to the high-dose spironolactone group will receive oral spironolactone (≥100 mg) on top of standard of care treatment for acute heart failure immediately after randomization and in the afternoon of each subsequent day unless the serum potassium level is >5 mmol/L. The exact dose will be determined based on a pre-specified algorithm provided.
  Other Names: Aldactone
  Arms: High-dose spironolactone

SUMMARY:
This is a prospective, single-center, open-label and randomized trial for evaluation of the effect of a 5-day administration of high doses of spironolactone (≥100mg daily) on diuresis, natriuresis, weight loss and levels of NT-proBNP in hospitalized patients with acute decompensated heart failure (ADHF). Mineralocorticoid receptor antagonists (MRAs) are recommended as standard of care (SOC) in management of heart failure (HF) patients. However, recommended doses of MRAs (up to 50mg daily) have any impact on signs and symptoms of volume overload. Therefore, the proposed study will aim to show the impact of high doses of spironolactone to improve diuresis, natriuresis, weight loss and levels of NT-proBNP in hospitalized patients with ADHF.

DETAILED DESCRIPTION:
Congestion represents a hallmark feature of ADHF, which is present in more than 90% of patients hospitalized for this diagnosis. Intravenous loop diuretics are the mainstay of treatment. Nonetheless, nearly half of the patients who are hospitalized for AdHF continue to have residual symptoms and sign of congestion at time of discharge. Various pharmacological and non-pharmacological interventions have been proposed over the past years as potential means for relieving congestion in hospitalized ADHF patients. However, their efficacy has not been shown.

Given that hyperaldosteronism is a key feature in HF, the hypothesis that administration of high doses of spironolactone can potentiate the natriuretic effects of loop diuretics and relieve congestion in the setting of ADHF has been raised.

According to the most recent guidelines spironolactone can be considered in combination with loop diuretic in patients with resistant edema or insufficient symptomatic response. However, spironolactone at a dose of 100 mg daily has failed to increase diuresis in patients with ADHF.

The present study will assess the effect of high per os doses of spironolactone (≥100mg) on top of SOC treatment compared with SOC treatment alone on diuresis, natriuresis, weight loss and levels of NT-proBNP in hospitalized patients with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute heart failure within the past 8 hours
* Two of the following: 1. edema, 2. ascites, 3. jugular vein distention, 4. pulmonary congestion
* NT-proBNP >1,000 pg/ml or >3,000 pg/ml (in the presence of atrial fibrillation)
* Per os mean daily loop diuretic dose equivalent to 80 mg of furosemide for at least 1 month prior to presentation and at least one of the following: 1. serum urea/serum creatinine > 50 at presentation, 2. serum creatinine increased >0.3 mg/dl compared with previous value (within the last year), 3. serum creatinine > 1.8 mg/dl.

Exclusion Criteria:

* pregnancy or breast feeding
* current acute coronary syndrome
* significant valvular disease
* pulmonary embolism
* allergy or intolerance to spironolactone
* current mechanical circulatory support
* primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy
* mean arterial pressure <65mmHg or systolic arterial pressure <90 mmHg at presentation
* anticipated use of inotropes or vasodilators (other than renal doses of dopamine, i.e. <2.5 μg/kg/min)
* anticipated need of ultrafiltration
* exposure to nephrotoxic agents within 3 days of presentation
* serum potassium> 5 mmol/L
* per os receipt of spironolactone or eplerenone in a dose > 50 mg daily prior to presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Daily urine output | 5 days
  Urine output in liters per 24 hours will be tracked from enrollment to day 5.

SECONDARY OUTCOMES:
Total urine output | 5 days
  Urine output in total liters from enrollment to day 5 will be measured.
Total weight change | 5 days
  Patient weight in kilos will be tracked from enrollment to day 5.
Daily weight change | 5 days
  Patient weight in kilos will be tracked from enrollment to day 5.
Natriuresis on days 1, 3 and 5 | 5 days
  Urine sodium will be measured on days 1, 3 and 5
Changes in natriuresis between days 1, 3 and 5 | 5 days
  Urine sodium will be measured on days 1, 3 and 5
Changes in NT-proBNP between days 1 and 5 | 5 days
  NT-proBNP will be measured on days 1, 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: John Barbetseas, MD, Study Chair — Laikon General Hospital
Locations (1):
- Laiko General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
The individual participant data of the study will be shared on reasonable request to the principle investigator

REFERENCES:
- [Background] Kapelios CJ, Bonou M, Vogiatzi P, Tzanis G, Mantzouratou P, Lund LH, Barbetseas J. Association Between High-Dose Spironolactone and Decongestion in Patients with Acute Heart Failure: An Observational Retrospective Study. Am J Cardiovasc Drugs. 2018 Oct;18(5):415-422. doi: 10.1007/s40256-018-0290-3. PMID 29971596